CLINICAL TRIAL: NCT03202264
Title: Team Approach to Polypharmacy Reduction to Improve Mobility (TAPER-Mobility): A Pilot Feasibility Study in a Long-Term Care Setting
Brief Title: Team Approach to Polypharmacy Reduction to Improve Mobility Long-Term Care
Status: Terminated | Type: Observational
Why Stopped: Difficulty with recruitment and staff retention.
Sponsor: McMaster University (Other)
Collaborators: The Labarge Optimal Aging Initiative (Other)
Responsible Party: Sponsor
Other Study IDs: TAPER-Mobility
Record Dates: First submitted 2017-02-23; First posted 2017-06-28 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Multi-morbidity; Medication Therapy Management; Polypharmacy
Keywords: Polypharmacy; Mobility; Multimorbidity; Drug Discontinuation; Patient Preference; eHealth
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAPERMD: 80 Long term care residents on 5 or more medications aged over 70 from 2 long term care facilities
  Interventions: Other: TAPER

INTERVENTIONS:
Other: TAPER — The intervention is medication reduction. This arm is comprised of:
  * Medication reconciliation
  * Identification of patient priorities for care
  * Identification of medications that are potentially appropriate for discontinuation/dose reduction
  * Linked pharmacist/family physician consultations with patient to discuss medication with intention to reduce
  * Identification of medications for trial of discontinuation/dose reduction (shared decision making)
  * Pause of medication and clinical monitoring

SUMMARY:
Medication side effects and interactions between medications are very common in older adults and are related to negative health outcomes, including mobility. In this study, the investigators will test a new process aimed at reducing unnecessary medication use and drug side effects in seniors using the best medical evidence and patient preferences for treatment. This study will assess how feasible the implementation of this intervention is within a long-term care facility as well as if it is possible. The study will also assess for any signals of reversal of medications related mobility impairments to reduce medications-related mobility impairment (fatigue, pain, falls) using the intervention. Participants in two long-term care facilities will participate in this study. Measures will include feasibility outcomes regarding the logistics of the intervention as well as patients outcomes (falls, hospitalizations, and medications) collected before and after implementation. Findings will inform the design of a randomized controlled trial to test the effect of this intervention on health outcomes.

DETAILED DESCRIPTION:
There are substantial associations between polypharmacy and reduced function from older adults and this is likely to be important in frail older adults both in long term care and in the community. The reversibility of drug-induced mobility impairment is unclear therefore the investigators plan to investigate signals of any impact of reducing polypharmacy on mobility. The investigators chose the long-term care setting given the presence of complete medication administration records and this patient population's high prevalence of polypharmacy and risk of adverse drug events. TAPERMD is an electronic tool for systematic medication reduction that incorporates patient priorities, electronic screening for potentially harmful medicines, supporting evidence tools and a monitoring pathway to support medication reduction. This study will examine the feasibility of this tool in a long-term care setting as well as examine. Participants in two long-term care facilities will participate in this study. Measures will include feasibility outcomes regarding the logistics of the intervention as well as patients outcomes (falls, hospitalizations, and medications) collected before and after implementation. Findings will inform a randomized controlled trial to measure the effect of this intervention on health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* residing in 2 long-term care facilities in Brampton, ON
* on 5 or more medications
* 70 years of age or older
* adequate English language

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults, 70 years of age or older, residing in 2 long-term care facilities located in the Brampton, Ontario, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be available on request to the Principal investigator. The data set will be uploaded as required for publication.

RESULTS

PARTICIPANT FLOW:
Groups:
- TAPERMD: 80 Long term care residents on 5 or more medications aged over 70 from 2 long term care facilities
  TAPER: The intervention is medication reduction. This arm is comprised of:
  * Medication reconciliation
  * Identification of patient priorities for care
  * Identification of medications that are potentially appropriate for discontinuation/dose reduction
  * Linked pharmacist/family physician consultations with patient to discuss medication with intention to reduce
  * Identification of medications for trial of discontinuation/dose reduction (shared decision making)
  * Pause of medication and clinical monitoring
Period: Overall Study
Arm/Group | TAPERMD
Started | 30
Completed | 14
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | TAPERMD
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two participants died prior to data collection.
  years
    number analyzed (Participants) | 28
    (all) | 90 (6.94)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two participants died prior to data collection.
  Participants
    number analyzed (Participants) | 28
    Female | 21
    Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  Canada | 30

OUTCOME MEASURES:

1. Primary Outcome: Successful Discontinuation (Difference in Mean Number of Medications; Reduction in Dose)
Description: Difference in mean number of medications; number of medications reduced in dose
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Medications Changed
Arm/Group | TAPERMD
Number analyzed (Participants) | 30
Medications Changed | 2.43 (2.98)

2. Secondary Outcome: Mobility-related Fatigue
Description: Avlund Mob-T Scale
Time Frame: Baseline, 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Level of Physical Functioning
Description: Manty survey
Time Frame: Baseline, 6 Months
Reporting Status: Not Posted

4. Secondary Outcome: Pain
Description: Brief Pain Inventory
Time Frame: Baseline, 6 Months
Reporting Status: Not Posted

5. Secondary Outcome: Falls
Description: Total count of falls recorded in hospital admissions, primary care records and patient report
Time Frame: Baseline, 6 Months
Reporting Status: Not Posted

6. Secondary Outcome: Sleep
Description: Pittsburgh Sleep Quality Index
Time Frame: Baseline, 6 Months
Reporting Status: Not Posted

7. Secondary Outcome: Decrease in Medication Side Effects and Symptoms
Description: Patient self-report change in symptoms, side effects, health improvements and problems
Time Frame: 1-week, 3-month, 6-month
Reporting Status: Not Posted

8. Secondary Outcome: Serious Adverse Events
Description: Any event that requires in-patient hospitalization or prolongation of existing hospitalization, causes congenital malformation, results in persistent or significant disability or incapacity, is life-threatening or results in death (Health Canada (2011) Guidance Document for Industry - Reporting Adverse Reactions to Marketed Health Products)
Time Frame: 1-week, 3-month, 6-month
Reporting Status: Not Posted

9. Secondary Outcome: Quality of Life
Description: EQ5D-5L
Time Frame: Baseline, 6-months
Reporting Status: Not Posted

10. Secondary Outcome: Physical Functioning Performance
Description: Timed-up and go Test
Time Frame: Baseline, 6-months
Reporting Status: Not Posted

11. Secondary Outcome: Physical Functioning Performance
Description: Timed 8-foot walk test
Time Frame: Baseline, 6-months
Reporting Status: Not Posted

12. Secondary Outcome: Performance of Activities of Daily Living
Description: Barthel Index
Time Frame: Baseline, 6-months
Reporting Status: Not Posted

13. Secondary Outcome: Strength
Description: Hand grip
Time Frame: Baseline, 6-months
Reporting Status: Not Posted

14. Secondary Outcome: Functional Ability
Description: Functional ability scale for the elderly
Time Frame: Baseline, 6-months
Reporting Status: Not Posted

15. Secondary Outcome: Healthcare Utilization
Description: Cost of hospitalizations
Time Frame: Baseline, 6-months
Reporting Status: Not Posted

16. Secondary Outcome: Healthcare Utilization
Description: Count of Emergency room visits
Time Frame: Baseline, 6-months
Reporting Status: Not Posted

17. Secondary Outcome: Healthcare Utilization
Description: Number of clinic visits
Time Frame: Baseline, 6-months
Reporting Status: Not Posted

18. Secondary Outcome: Feasibility Outcomes
Description: Number of participants that refuse recruitment
Time Frame: 6 months
Reporting Status: Not Posted

19. Secondary Outcome: Feasibility Outcomes
Description: Retention rates
Time Frame: 6 months
Reporting Status: Not Posted

20. Secondary Outcome: Feasibility Outcomes
Description: number of canceled appointments
Time Frame: Baseline, 6 months
Reporting Status: Not Posted

21. Secondary Outcome: Feasibility Outcomes
Description: Time to complete measures
Time Frame: Baseline, 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months from Physician Visit to Follow-up.
Description: Events were recorded via patient chart audit.
Arm/Group | TAPERMD
All-Cause Mortality (participants affected / at risk) | 8/30
Serious Adverse Events (participants affected / at risk) | 5/30
Other Adverse Events (participants affected / at risk) | 14/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAPERMD (N=30)
AECOPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
decreased level of consciousness (Nervous system disorders) | 2 (2)
vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
wound infested with maggots (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAPERMD (N=30)
Fall resulting in no or minor injury (Injury, poisoning and procedural complications) | 9 (16)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tooth extraction & complications (Injury, poisoning and procedural complications) | 2 (4)
large skin tear/pressure ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
diagnosed with diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
worsening of Parkinson's Disease with dementia (Nervous system disorders) | 1 (1)
increased leg edema (Cardiac disorders) | 1 (1) — History of congestive heart failure
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT03202264/Prot_SAP_000.pdf